CLINICAL TRIAL: NCT01177462
Title: The Transformation of Coordinates Between Somatosensory and Visual Systems: a Neurophysiological Study
Brief Title: Transformation of Somatosensory and Visual Coordinate Systems
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Cheng Pei, Attending Physician, Chang Gung Memorial Hospital
Other Study IDs: CMRPG590021G
Record Dates: First submitted 2010-07-29; First posted 2010-08-09 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Stroke
Keywords: coordinate system; normal
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- hemineglect stroke patients: Stroke patients with hemineglect
- Control stroke patients: Stroke patients without hemineglect
- Normal control: Normal subjects

SUMMARY:
Manipulation of object is a multisensory experience that includes tactile motion between the object and the fingerpad, visual motion elicited by the motion the object and the movement of the hand, and the active motor commend to control upper limb and hand conformation. It remains to be determined how such a complex interaction between touch and vision could be achieved effortlessly. In the present study, we will investigate how the motion information is transformed between touch and vision using the most novel approaches in human psychophysics, neuropsychology and monkey neurophysiology. Specifically, we will present tactile motion on primate fingerpads using a recently developed ball stimulator with a design in which we vary the direction of motion with respect to the skin surface and also vary the hand conformation and position. This setup allows us to systematically sample the possible scenarios involving coordinate transformation between the somatosensory and visual systems in conditions that could occur in hand exploration and object manipulation in daily life. We will present these tactile stimuli on normal human subject as well as stroke patients such as patients with spatial hemineglect. Finally, we will record from macaque monkeys in cortical areas that are thought to underlie the transformation of coordinates, such as the primary somatosensory cortex and posterior parietal cortex. The results of the present study will contribute to the understanding of multisensory integration and the rehabilitation for patients with impaired use of spatial information.

ELIGIBILITY:
For stoke patients

Inclusion Criteria:

* stroke patients
* stable medical condition
* can cooperate in evaluation

Exclusion Criteria:

* peripheral neuropathy
* limb ambulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit 40 normal healthy adult subjects (equal to and more than 18 years old); the exclusion criteria are subjects with brain pathology, peripheral neuropathy and limb amputation. We will also recruit 50 stroke patients, the including criteria are stroke patients with stable medical condition and being capable of receiving the evaluations. In this group, stroke patients with peripheral neuropathy, and unstable medical condition.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Perceived direction of tactile motion | Once; specifically for stroke patients, 6 months after the onset of stroke
  Detail description for time frame of assessment:
  (1) for stroke patients, the assessment will be performed "in average" 6 months after the onset of stroke (2) for normal subjects: assessment will be done when the subject is willing to participate (3) the subject might come to the lab more than once if the experiment can not be completed in one session
  Assessment:
  We present tactile motion using tactile stimulators to (1)different digits (2)different hand conformations and (3) different hand positions relative to the trunk

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Cheng Pei, MD PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan, Taiwan